CLINICAL TRIAL: NCT04467346
Title: Bioequivalence Study Between Temozolomide Oral Suspension (Ped-TMZ) and Temodal® Capsules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orphelia Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ORP-TMZ-I-a
Record Dates: First submitted 2020-03-27; First posted 2020-07-13 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Therapeutic Equivalency

STUDY DESIGN:
Intervention Model Description: The study is an open label, randomized, crossover, 2-period study in 30 male/female patients with primary CNS malignancies. Patients will receive, under fasting conditions, 200 mg/m² of Temozolomide Oral Suspension (Ped-TMZ) or Temodal®, as single oral administration in 2 different study periods depending on the randomization, with no wash out period between administrations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ped-TMZ (Experimental): Single oral administration on D1 or D2 according to randomization at the dose of 200 mg/m2. Ped-TMZ will be administered using the provided dosing oral syringes and followed by a glass of 240 ml of water (for mouth rinsing) in sitting position and under fasting condition.
  Interventions: Drug: Ped-TMZ
- Temodal capsule (Active Comparator): Single oral administration on D1 or D2 according to randomization at the dose of 200 mg/m2. The administration will take place around 8:00 a.m. followed with 240 mL of tap water, in sitting position and under fasting condition
  Interventions: Drug: Ped-TMZ

INTERVENTIONS:
Drug: Ped-TMZ — Ped-TMZ will be administered using the provided dosing oral syringes and followed by a glass of 240 ml of water (for mouth rinsing) in sitting position and under fasting condition for at least 8 hours before dosing
  Other Names: Temozolomide Oral Suspension

SUMMARY:
Primary objective:

• Evaluate bioequivalence between Temozolomide Oral Suspension and Temodal® capsules for oral administration.

Secondary objectives:

* Define the pharmacokinetic parameters of Temozolomide Oral Suspension.
* Assess the buccal safety of Temozolomide Oral Suspension.

DETAILED DESCRIPTION:
The study is an open label, randomized, crossover, 2-period study in 30 male/female patients with primary CNS malignancies. Patients will receive, under fasting conditions, 200 mg/m² of Temozolomide Oral Suspension (Ped-TMZ) or Temodal®, as single oral administration in 2 different study periods depending on the randomization, with no wash out period between administrations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed glioblastoma multiforme treated with temozolomide (200mg/m2) as monotherapy and patients with recurrent or progressive malignant glioma treated with temozolomide as monotherapy (200mg/m2).
* Male and female patients at least 18 of age.
* Non-pregnant, non-breast feeding female.
* Body mass index (weight/height²) in the range of 18.5 to 30 kg/m².
* Having given a written informed consent

Exclusion Criteria:

* Co-administration of sodium valproate
* Patients with (naso)gastric tubes
* Patients receiving 150 mg/m² and not eligible to the 200 mg/m² dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Primary pharmacokinetic parameter: Cmax | Day 1 or Day 2
  The Cmax pharmacokinetic parameter will be determined from temozolomide plasma concentrations
Primary pharmacokinetic parameter: AUC0-t | Day 1 or Day 2
  The AUC0-t pharmacokinetic parameter will be determined from temozolomide plasma concentrations

SECONDARY OUTCOMES:
Secondary pharmacokinetic parameter: AUC0-inf | Day 1 or Day 2
  The AUC0-inf pharmacokinetic parameter will be determined from temozolomide plasma concentrations
Secondary pharmacokinetic parameter: tmax | Day 1 and Day 2
  The tmax pharmacokinetic parameter will be determined from temozolomide plasma concentrations
Secondary pharmacokinetic parameter: λ | Day 1 and Day 2
  The λ pharmacokinetic parameter will be determined from temozolomide plasma concentrations
Secondary pharmacokinetic parameter: t1/2 | Day 1 and Day 2
  The t1/2 pharmacokinetic parameters will be determined from temozolomide plasma concentrations
Secondary pharmacokinetic parameter: residual area | Day 1 and Day 2
  The residual area of temozolomide will be determined from temozolomide plasma concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Lemarchand, PharmD, Study Director — Orphelia Pharma
Locations (3):
- France (3):
  - Service de neuro-oncologie - Hospices Civils de Lyon, Bron, Rhône
  - CHU de Bordeaux, Bordeaux
  - Hôpital de la Timone (AP-HM), Marseille

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ducray F, Ramirez C, Robert M, Fontanilles M, Bronnimann C, Chinot O, Estrade F, Durando X, Cartalat S, Bastid J, Bienayme H, Lemarchand C. A Multicenter Randomized Bioequivalence Study of a Novel Ready-to-Use Temozolomide Oral Suspension vs. Temozolomide Capsules. Pharmaceutics. 2023 Nov 24;15(12):2664. doi: 10.3390/pharmaceutics15122664. PMID 38140005